CLINICAL TRIAL: NCT01668992
Title: Impact Evaluation of a Family-based Intervention With Burmese Migrant and Displaced Children and Families in Tak Province, Thailand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Rescue Committee (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Harvard School of Public Health (HSPH) (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21050
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Parenting Practices; Family Functioning; Child Psychosocial Well-being; Alcohol Use
Keywords: Parenting; Discipline; Family interventions; Thailand; Migration
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family intervention (Experimental): Families receive 12-week program on parenting skills, discipline methods and family communication.
  Interventions: Behavioral: Family intervention
- Waitlist control (No Intervention): Families are on a waitlist and receive the intervention only after the trial is complete.

INTERVENTIONS:
Behavioral: Family intervention — 12-week parenting skills program for Burmese migrant and displaced children and families.
  Other Names: Happy Families Program
  Arms: Family intervention

SUMMARY:
The study will evaluate the impact of a family-based intervention on the well-being of Burmese migrant and displaced children and families living in Tak province, Thailand. The methodology used in the impact evaluation study is a randomized waitlist controlled trial.

The study hypothesizes that participation in a family-based intervention will lead to improved parenting practices and child and family outcomes, as follows.

Primary hypotheses:

1. Parents/caregivers participating in the family-based intervention will report increased knowledge and use of positive parenting skills compared to control;
2. Parents/caregivers participating in the family-based intervention will report less use of physical punishment and other harsh forms of discipline compared to control;
3. Parents/caregivers and children participating in the family-based intervention will report higher levels of family functioning and cohesion compared to control.

Secondary hypotheses:

1. Parents/caregivers and children participating in the family-based intervention will report lower levels of externalizing and internalizing child behaviors compared to control;
2. Parents/caregivers and children participating in the family-based intervention will report higher levels of child resilience and psychosocial well-being compared to control;
3. Parents/caregivers participating in the family-based intervention will report lower levels of alcohol use compared to control.

ELIGIBILITY:
Inclusion Criteria:

* Of Burmese origin
* Currently living in one of 20 target communities in Tak province, Thailand
* Primary caregiver to at least one child aged 8 to 12 years
* Child aged 8 to 12 years
* Participating in the family intervention

Exclusion Criteria:

* Children living in orphanages, boarding houses, factories or other institutions
* Persons with severe cognitive or physical disability who are impaired and unable to understand and give informed consent

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 992 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Parenting practices | One month and six months post-intervention
  Changes in knowledge and use of positive parenting skills; change in use of physical punishment and other harsh forms of discipline.

SECONDARY OUTCOMES:
Child psychosocial well-being | One month and six months post-intervention
  Changes in report of child externalizing and internalizing symptoms and resilience.

OTHER OUTCOMES:
Family functioning and cohesion | One month and six months post-intervention
  Changes in levels of family communication, decision-making and relationships.
Alcohol use | One month and six months post-intervention
  Changes in adult alcohol use.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa S Betancourt, Sc.D., M.A., Principal Investigator — Harvard School of Public Health (HSPH); Jeannie Annan, PhD, Principal Investigator — International Rescue Committee
Locations (1):
- International Rescue Committee (IRC) Thailand, Mae Sot, Changwat Tak, Thailand

REFERENCES:
- [Derived] Puffer ES, Annan J, Sim AL, Salhi C, Betancourt TS. The impact of a family skills training intervention among Burmese migrant families in Thailand: A randomized controlled trial. PLoS One. 2017 Mar 28;12(3):e0172611. doi: 10.1371/journal.pone.0172611. eCollection 2017. PMID 28350809